CLINICAL TRIAL: NCT06440005
Title: A Phase 1, Open-Label, Dose-Escalation and Expansion Study of AGX101, a TM4SF1 Directed Antibody Drug Conjugate in Patients With Unresectable, Locally Advanced, or Metastatic Solid Tumors
Brief Title: A Study to Evaluate Safety, Tolerability and Preliminary Activity of AGX101 in Participants With Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Angiex, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: AGX101-001
Record Dates: First submitted 2024-05-26; First posted 2024-06-03 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Cancer; Advanced Cancer; Locally Advanced Carcinoma; Metastatic Solid Tumor; Breast Cancer; Prostate Cancer; Colorectal Cancer; Pancreatic Cancer; Liver Cancer; Angiosarcoma; Solid Tumor
Keywords: ADC; Antibody Drug Conjugate; AGX101
MeSH Terms: conditions — Neoplasms; Neoplasm Metastasis; Breast Neoplasms; Prostatic Neoplasms; Colorectal Neoplasms; Pancreatic Neoplasms; Liver Neoplasms; Hemangiosarcoma

STUDY DESIGN:
Intervention Model Description: A mTPI-2 design (Guo et al, 2017) with a target DLT rate of at most 30% will be applied for dose-escalation and expansion to determine the AGX101 RP2D.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Dose Escalation Phase (Experimental): AGX-101, initial 90-minute IV infusion, second 60-minute IV infusion and 30 minute subsequent IV infusions on Day 1 of every 3, 6 or 9-week cycle in Dose Escalation Phase. Dose escalation will be carried out in sequential cohorts of escalating doses, with an expansion cohort in advanced angiosarcoma.
  Interventions: Drug: AGX101
- Dose Expansion Phase (Experimental): AGX-101, initial 90-minute IV infusion, second 60-minute IV infusion and 30 minute subsequent IV infusions on Day 1 of every every 3, 6 or 9-week cycle in Dose Escalation Phase. Dose expansion will be carried out with a selected dose and selected cancer type.
  Interventions: Drug: AGX101

INTERVENTIONS:
Drug: AGX101 — Antibody Drug Conjugate
  Other Names: ADC

SUMMARY:
AGX101 is an antibody-drug conjugate (ADC) therapy for tumor-forming cancers. The purpose of this study is to learn about AGX101 effects and safety at various dose levels in an all-comers advanced solid cancer patient population. AGX101will be administered intravenously.

Dosing of AGX101 will be repeated once every 3, 6 or 9 weeks. Participants may continue study treatment until disease progression, unacceptable toxicity, or consent withdrawal. Subjects will attend an end of treatment visit and will receive two safety follow-up telephone contacts up to 90 days following the last dose of study drug.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed unresectable, locally advanced, or metastatic solid tumors.
* Refractory to or relapsed after all standard therapies known to provide proven clinical benefit, unless the patient is not a candidate for standard treatment, there is no standard treatment, or the patient refuses standard treatment after expressing an understanding of all available therapies with proven clinical benefit
* Willing to authorize use of existing archival tissue, unless otherwise discussed with Sponsor
* Time since the last dose of prior therapy to treat underlying malignancy (including other investigational therapy): Systemic cytotoxic chemotherapy: ≥ the duration of the most recent cycle of the previous regimen (with a minimum of 2 weeks for all, except 6 weeks for systemic nitrosourea or systemic mitomycin-C); Biologic therapy (eg, antibodies): ≥ 3 weeks; Small molecule therapies: ≥ 5 × half-life
* Have an ECOG performance status of 0 to 1
* Have adequate organ function
* LVEF ≥ 50%, as determined on cardiac ECHO or cardiac multiple-gated acquisition (MUGA) scan
* Highly effective contraception for both male and female patients throughout the study

Exclusion Criteria:

* Colorectal cancer patients with an unresected primary colorectal tumor and non-small-cell lung cancer with predominant squamous histology (ie, squamous cell carcinoma of the lung) are excluded unless otherwise discussed and approved by Sponsor
* Clinically unstable central nervous system (CNS) tumors or brain metastasis (stable and/or asymptomatic CNS metastases allowed)
* Have not recovered to ≤ Grade 1 or baseline from all AEs due to previous therapies (patients with ≤ Grade 2 neuropathy, endocrine-related irAEs, or other AEs may be eligible after discussion with the Sponsor)
* Has an active vasculitis that has required systemic treatment in the past 2 years prior to starting study treatment
* Significant (ie, ≥ Grade 2) ocular disturbances
* Variceal bleeding within 6 months prior to treatment, currently untreated or incompletely treated varices with bleeding, or who otherwise are at a high risk of bleeding
* Any other concurrent antineoplastic treatment except for allowed local radiation of lesions for palliation (to be considered non-target lesions after treatment) and hormone ablation
* Uncontrolled or life-threatening symptomatic concomitant disease, including known symptomatic HIV positive with an AIDS defining opportunistic infection within the last year, known symptomatic active hepatitis B or C, or known active tuberculosis
* Has undergone a major surgery within 3 weeks prior to starting study treatment or has inadequate healing or recovery from complications of surgery prior to starting study treatment
* Has received prior radiotherapy within 2 weeks prior to starting study treatment
* Has or had a potentially life-threatening second malignancy requiring systemic treatment within the last 3 years, or which would impede evaluation of treatment response
* Clinically significant cardiovascular disease
* Patients on a potent CYP3A inhibitor or CPY3A inducer who cannot be changed to another medication
* Has an active infection requiring concurrent systemic antibiotic therapy
* A woman of child-bearing potential (WOCBP) who has a positive pregnancy test prior to treatment
* Is breastfeeding or expecting to conceive or father children within the projected duration of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-07-22 (Actual); Primary Completion 2026-09-06 (Estimated); Study Completion 2027-09-06 (Estimated)

PRIMARY OUTCOMES:
Acceptable maximum tolerated dose for participants | 21 days following the first dose of AGX101 (Day 1 through Day 21)
  Maximum tolerated dose (MTD) and the dose-limiting toxicities (DLTs) of AGX101 will be characterized
Number of participants with adverse events | Screening through end of treatment, approximately 6 months and up to 3 years
  Evaluation of the incidence, severity, and duration of adverse events

SECONDARY OUTCOMES:
Terminal elimination half life (PK) | 22 days following the first dose of AGX101 (Day 1 through Day 22)
  Determination of the terminal elimination half-life (t½)
AUC (PK) | 22 days following the first dose of AGX101 (Day 1 through Day 22)
  Determination of the AUC in 1 dosing interval
Cmax (PK) | 22 days following the first dose of AGX101 (Day 1 through Day 22)
  Determination of the Cmax concentration over a dosing interval, systemic clearance, volume of distribution at steady-state (Vss), and accumulation ratio from first dose to steady-state
Number of Participants with Antidrug Antibodies (ADA) to AGX101 | Approximately 6 months and up to 3 years
  Incidence and titers of ADA will be measured
Efficacy as measured by Proportion of Participants with Objective Response Rate (ORR) According to RECIST v1.1 Evaluated by the Investigator | Approximately 6 months and up to 3 years
  Determination the objective response rate (ORR)
Efficacy as measured by Duration of Response (DoR) Assessed by Investigator | Approximately 6 months and up to 3 years
  Determination of the duration of response (DoR)
Efficacy as measured by Disease Control Rate (DCR) | Approximately 6 months and up to 3 years
  Determination of the disease control rate (DCR)
Efficacy as measured by Proportion of Participants with Progression Free Survival (PFS) According to RECIST v1.1 Evaluated by the Investigator | Approximately 6 months and up to 3 years
  Determine progression-free survival (PFS)/PFS assessed per immune-related response evaluation criteria (iPFS).
Efficacy as measured by Duration of Treatment | Approximately 6 months and up to 3 years
Overall Survival | Approximately 6 months and up to 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Glen Weiss, MD, Study Director — Medical Lead
Locations (6):
- United States (6):
  - USC/Norris Comprehensive Cancer Center, Los Angeles, California
  - Florida Cancer Specialist, Sarasota, Florida
  - Washington University School of Medicine, St Louis, Missouri
  - Sarah Cannon Research Center, Nashville, Tennessee
  - NEXT Oncology, San Antonio, Texas
  - NEXT Oncology, Fairfax, Virginia